CLINICAL TRIAL: NCT03933761
Title: A Phase II, Signal-Seeking Trial of the Clinical Benefit Rate Associated With Pamiparib in Subjects With Germline or Somatic BRCA1/2 High Grade Serous Ovarian Cancer or Carcinosarcoma Who Have Progressed on P-gp Substrate Chemotherapy or PARPi With the Presence of an ABCB1 Fusion and the Absence of a BRCA1/2 Reversion
Brief Title: Pamiparib in Fusion Positive, Reversion Negative High Grade Serous Ovarian Cancer or Carcinosarcoma With BRCA1/2 Gene Mutations If Progression on Substrate Poly ADP Ribose Polymerase Inhibitbor (PARPI) or Chemotherapy
Acronym: PRECISE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No eligible patient identified after 18 evaluable patients underwent pre-screening over a 2 year period.
Sponsor: Australia New Zealand Gynaecological Oncology Group (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZGOG 1721/2018
Record Dates: First submitted 2019-04-02; First posted 2019-05-01 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Cancer; Carcinosarcoma
Keywords: High grade serous; ABCB1 fusion positive; BRCA 1/2 reversion negative; Platinum resistant; Platinum sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Carcinosarcoma | interventions — pamiparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pamiparib (BGB-290) (Experimental): Drug: Pamiparib Oral capsules 60mg twice daily continuously Although treatment is continuous, a cycle is defined as 4 weeks or 28 days.
  Interventions: Drug: Pamiparib

INTERVENTIONS:
Drug: Pamiparib — 60 mg of pamiparib (3 capsules of 20mg) will be administered orally twice a day, once in the morning and once in the evening continuously in 28 day cycles.
  Other Names: BGB-290

SUMMARY:
This study is a phase II, multi-centre, open label study in patients with advanced ovarian cancer. The treatment being tested is Pamiparib, with daily dosing.

All patients enrolled to the study will receive treatment with pamiparib. Patients will be selected for entry into the study based on the molecular signature of their cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the deadliest gynaecologic cancer in Western women. Although initially responsive to therapy, drug resistance commonly evolves.

Novel mechanisms of drug resistance in ovarian cancer have been identified and include genetic mutations that result in the activation of a drug efflux pump and secondary mutations in BRCA1/2 genes that restore the cancer cell's ability to repair treatment related DNA damage. It is hypothesized that patients with BRCA1/2 mutant high grade serous ovarian cancer or carcinosarcoma who have progressed on recent therapy and have an activated efflux pump without a secondary BRCA1/1 mutation will be selectively sensitive to a new PARPi, Pamiparib, which does not get effluxed out of cancer cells.

The primary objective of this trial is to assess the clinical benefit rate at > 4 months in 2 cohorts of patients (cohort 1: post substrate-PARP inhibitor and cohort 2: post chemotherapy) defined as response or absence of progression. Secondary objectives are to determine the median progression free and overall survival of patients treated with Pamiparib and the impact on symptom burden and benefit.

ELIGIBILITY:
Inclusion Criteria - Pre-Screening

1. Patient has provided written informed consent for pre-screening
2. Patient is able to comply with the study protocol and follow-up procedures, in the Investigator's judgement
3. Patient is female aged ≥ 18 years at time of consent
4. ECOG performance status 0-2 (refer to Appendix 1)
5. Patient has the ability to take oral medications without medical history of malabsorption or other chronic gastrointestinal disease, or other conditions that may harm compliance and/or absorption of the study agent
6. Patients with a histopathological diagnosis of HGSC or carcinosarcoma of the ovary (including primary peritoneal cancers and fallopian tube cancers) as defined by histological diagnosis and immunohistochemistry (IHC) and with a germline or somatic BRCA1/2 mutation:

   * Mixed histologies are allowed provided that >80% of the primary tumour is a HGSC based on diagnostic pathology review and IHC profile
7. Patients with progressive disease defined by GCIG CA-125 and/or RECIST v1.1 criteria after 3 or more lines of chemotherapy or after progression on a P-gp substrate PARPi (i.e.

   olaparib, niraparib)
   * Patients may continue on treatment as per standard of care by their usual clinician while awaiting the results of pre-screening with no impact on usual care
   * Patients who have been treated with both substrate PARPi and substrate chemotherapy will be considered eligible for either cohort 1 or cohort 2 based on the therapy they have most recently progressed on (cohort 1 is progression on PARPi and cohort 2 is progression on chemotherapy)
8. Disease that is amenable to a biopsy and/or ascitic drainage

   * Lesions intended to be biopsied should not be target lesions with the preference of the biopsy site having progressed on most recent imaging where clinically safe and feasible
9. Patient has a life expectancy > 12 weeks
10. Patient has consented to the collection and use of their fresh tumour biopsies and/or ascites samples

Exclusion Criteria - Pre-Screening

1. Patients with a clear cell, mucinous, or other non-high grade serous histological subtype
2. Prior treatment with non-substrate P-gp PARPi (pamiparib or veliparib)

   * Prior treatment with substrate PARPi is allowed (olaparib, niraparib, rucaparib, and talazoparib)
3. Patients who are pregnant or nursing
4. Patient has a diagnosis of myelodysplastic syndrome (MDS)
5. Patient has other diagnoses of malignancy

   * Except for surgically excised non-melanoma skin cancer, adequately treated carcinoma in situ of the cervix, adequately treated non-invasive bladder cancer, ductal carcinoma in situ treated surgically with curative intent, or a malignancy diagnosed >2 years ago with no current evidence of disease and no therapy ≤2 years prior to pre-screening
6. Prior radiation therapy to target lesions in the absence of documented progression at the treated target lesion
7. Patient has uncontrolled pleural effusion, pericardial effusion, or ascites requiring weekly recurrent drainage procedures
8. Known history of intolerance to the excipients of the pamiparib capsule
9. Active bleeding disorder, including gastrointestinal bleeding, as evidenced by hematemesis, significant hemoptysis, or melena ≤6 months prior to registration to pre-screening
10. Previous complete gastric resection, chronic diarrhea, active inflammatory gastrointestinal disease, or any other disease-causing malabsorption syndrome

    * Gastroesophageal reflux disease under treatment with proton-pump inhibitors is allowed

Inclusion Criteria - Main Study

1. Patient has provided written informed consent for main PRECISE study
2. Patient continues to meet all pre-screening inclusion criteria
3. Patient has an ABCB1 fusion(s) and the absence of a BRCA1/2 reversion
4. Patient has platinum sensitive or platinum resistant HGSC

   * Patients who are refractory (progress during or within 4 weeks) to second or subsequent lines of platinum-based chemotherapy are eligible
   * Patients who are primary platinum refractory (progress during or within 4 weeks of first line chemotherapy) are considered ineligible
5. Recurrent disease that is measurable according to RECIST v1.1 or evaluable disease using CA-125 according to GCIG criteria
6. Adequate haematologic and end-organ function, as defined by the following laboratory results (obtained within 7 days prior to registration to the main study):

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Haemoglobin (Hb) ≥ 90 g/L (≥ 28 days after transfusion)
   * Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2 by the Modification of Diet in Renal Disease study equation (MDRD STUDY EQ; www.mdrd.com or Appendix 5)
   * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * ≤ 4 x ULN, if Gilbert's syndrome or if indirect bilirubin concentrations suggestive of extrahepatic source of elevation
   * Aspartate and alanine aminotransferase (AST and ALT) ≤ 3 x upper limit of normal (ULN) or ≤ 5 x ULN for patients with liver metastases
7. Females who are of childbearing potential

   * Females of childbearing potential require a negative serum pregnancy test within 7 days prior to registration into the main study
8. Females of childbearing potential must practice highly effective methods of birth control (refer to Appendix 2) for the duration of the study and for at least 6 months after last study drug
9. Patients must have recovered to ≤ grade 1 from their treatment-related adverse event (AE) with the exception of alopecia and peripheral neuropathy
10. Able to provide a formalin-fixed paraffin embedded (FFPE) tumour block, representative of the patient's primary disease

    * In cases where there is insufficient FFPE tumour, a discussion with the Coordinating Principal Investigator (CPI) must be had before registration to the main study

Exclusion Criteria - Main Study

1. Patients who have received chemotherapy, biologic therapy, immunotherapy, investigational agent, anticancer Chinese medicine, or herbal remedies ≤ 5 half-lives if the half-life is known, ≤ 14 days if not known, prior to registration to the main study

   * Bisphosphonate and denosumab use are allowed on study, if administered at a stable dose > 28 days prior to registration to the main study
2. The use or anticipated need for food or drugs known to be strong CYP3A inducers (Appendix 7) ≤ 5 half-lives if the half-life is known or ≤ 14 days if not known prior to registration to the main study
3. Major surgical procedure, open biopsy, or significant traumatic injury ≤ 14 days prior to registration to the main study, or anticipation of need for major surgical procedure during the course of the study

   * Placement of vascular access device is not considered major surgery
4. Prior radiation therapy ≤ 14 days prior to registration to the main study to non-target lesions. Patients who have received palliative radiotherapy of non-target lesions for local symptom control > 14 days prior to registration to the main study must have stabilisation of any AEs or a return to baseline prior to registration to the main study
5. Leptomeningeal disease or uncontrolled, untreated brain metastases
6. Patients with a history of treated and asymptomatic brain metastases are eligible, provided they meet all of the following:

   * Only supratentorial metastases
   * Brain imaging at screening without evidence of interim progression
   * No ongoing requirement for corticosteroids as therapy for brain metastases
   * Anticonvulsants at a stable dose allowed (except for contraindicated medications carbamazepine and phenytoin)
   * No stereotactic radiation or whole-brain radiation ≤ 14 days prior to registration to the main study
7. Any of the following cardiovascular criteria:

   * Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days prior to registration to the main study
   * Symptomatic pulmonary embolism ≤ 28 days prior to registration to the main study
   * Any history of acute myocardial infarction ≤ 6 months prior to registration to the main study
   * Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV (refer to Appendix 8) ≤ 6 months prior to registration to the main study
   * Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months prior to registration to the main study
   * Any history of cerebrovascular accident (CVA) ≤ 6 months prior to registration to the main study
8. Active infection requiring systemic treatment, acute/viral hepatitis or active chronic hepatitis B or C or active tuberculosis

   * Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is > 500 IU/mL or patients with active hepatitis C should be excluded. Note: Inactive hepatitis B surface antigen carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL), and cured hepatitis C patients can be enrolled

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with high grade serous ovarian cancinoma or carcinosarcoma.
Enrollment: 0 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | Assessed at 16 weeks after commencing treatment.
  as assessed by RECIST v1.1 or by Gynaecological Cancer Intergroup (GCIG) Cancer antigen (CA)-125 criteria

SECONDARY OUTCOMES:
Frequency of ABCB1 fusions and BRCA1/2 reversions | At Baseline
  in patients with germline or somatic BRCA1/2 high grade serous cancer or carcinosarcoma
Median progression free survival | Through study completion, on average 6 months.
  in BRCA1/2 high grade serous cancer or carcinosarcoma patients with ABCB1 fusions in the absence of BRCA1/2 reversions treated with pamiparib.
Median overall survival | Assessed for up to 3 years after the last patient enrolled has commenced treatment.
  in BRCA1/2 high grade serous cancer or carcinosarcoma patients with ABCB1 fusions in the absence of BRCA1/2 reversions treated with pamiparib.
Duration of response | Assessed for up to 3 years after the last patient enrolled has commenced treatment.
  Duration of response according to RECIST v1.1 in the subset of patients who achieved partial response or complete response.
Best overall response according to RECIST v1.1 | Assessed for up to 3 years after the last patient enrolled has commenced treatment.
  Best overall response is the best response from commencement of treatment according to RECIST v1.1
Best overall response according to CA-125 | Assessed for up to 3 years after the last patient enrolled has commenced treatment.
  defined as best response from commencement of treatment determined by GCIG CA-125 criteria
Patient reported symptom burden | At the time of consent to screening, at every cycle to 16 weeks, then every 4 cycles, and again at the time of progression. Assessed for up to 3 years after the last patient enrolled has commenced treatment.
  Using the Measure of Ovarian Cancer Symptoms and Treatment Concerns (MOST) v2 patient reported outcome measure (PROM)
  * The scale measures disease or therapy related symptoms and symptom burden and well-being
  * Scale ranges: Subscales are reported in five different categories with the subscale score ranges below
    * Abdominal symptoms, higher values reflecting worst possible symptoms
    * Disease or treatment-related symptoms, higher values reflecting worst possible symptoms
    * Chemotherapy-related symptoms, higher values reflecting worst possible symptoms
    * Psychological symptoms, higher values reflecting worst possible symptoms
    * Well-being, higher values reflecting best possible symptoms
  * Each of the 5 subscales can be scored and analysed separately (item by item) or by taking the average of the component items.
Patient reported results of the 40 item State-trait anxiety inventory for adults (STAI-ADTM) | This will be assessed 3 times - at the time of pre-screening consent, immediately prior to clinician consult with notification of pre-screening results, and immediately following notification of pre-screening results.
  * The scale measures state level anxiety (S-Anxiety or current levels) and trait anxiety levels (T-anxiety or how someone generally feels)
  * Scale ranges: STA Form Y-1 includes 20 items/questions, with a total score range of 20-80, and STA Form Y-2 includes 20 items/questions, with a total score range of 20-80. Each scored item/question is then given a weighted score of 1 to 4 with a rating of 4 indicative of a high level of anxiety for 10 x S-Anxiety items and 11 x T-Anxiety items. A high rating indicates the absences of anxiety for the remaining 10 S-Anxiety items and 9 T-Anxiety items. The scoring weights for the anxiety-present items are the same as the chosen numbers on the form and the scoring weight for the anxiety-absent items are reversed.
  * For each form separately, weighted scores are then totalled and averaged. Groups of respondents will be identified (including most anxious, least anxious, and middle) based on top, bottom, and middle percentiles.
The type, grade and relationship to treatment of adverse events | During the treatment period, on average 3 years
  The type, grade and relationship to treatment of adverse events, assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alison Freimund, Principal Investigator — Peter MacCallum Cancer Centre, Australia

IPD SHARING:
Plan to Share IPD: No